CLINICAL TRIAL: NCT01345331
Title: Ear Electro-stimulation for Chronic Pelvic Pain
Acronym: RAVANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Dr. Vitaly Napadow, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2008p001019
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Stimulation (Experimental): Ear stimulation at specific points should work by stimulating a nerve called the vagus nerve. Previous research has shown that stimulating this nerve can help patients feel less pain.
  Interventions: Behavioral: Real stimulation VS Sham
- Sham (Sham Comparator): The sham treatment will use the same equipment as the real treatment, but the participant will not receive any real stimulation to the ear.
  Interventions: Behavioral: Real stimulation VS Sham

INTERVENTIONS:
Behavioral: Real stimulation VS Sham — Ear stimulation at specific points should work by stimulating a nerve called the vagus nerve. Previous research has shown that stimulating this nerve can help patients feel less pain. During any testing session, participants may receive either the real ear stimulation or a sham (placebo) treatment. The sham treatment will use the same equipment as the real treatment, but will not deliver any real stimulation to the ear. We use placebo/sham procedures in research to make sure that the study results are related to the study procedure, and not to other reasons.

SUMMARY:
The Brigham and Women's Pain Management Center is conducting a research study for chronic pelvic pain patients due to endometriosis. The study will assess the effect of electro-stimulation for the treatment of Chronic Pelvic Pain. You may be eligible if you have chronic pelvic pain due to endometriosis, are between the ages of 21- 64, and not taking opioid medication (such as morphine or oxycodone). The study will require two visits, each lasting about 2 hours. The study takes place at the Brigham & Women's Pain Management Center, 850 Boylston St., Chestnut Hill. Please contact Chrissie Cahalan at 617-732-9014 or ccahalan1@partners.org if interested.

DETAILED DESCRIPTION:
The Brigham and Women's Pain Management Center is conducting a research study for chronic pelvic pain patients due to endometriosis. The study will assess the effect of electro-stimulation for the treatment of Chronic Pelvic Pain. You may be eligible if you have chronic pelvic pain due to endometriosis, are between the ages of 21- 64, and not taking opioid medication (such as morphine or oxycodone). The study will require two visits, each lasting about 2 hours. The study takes place at the Brigham & Women's Pain Management Center, 850 Boylston St., Chestnut Hill. Please contact Chrissie Cahalan at 617-732-9014 or ccahalan1@partners.org if interested.

Vitaly Napadow, Ph.D., Lic.Ac. Assistant Professor Dept. of Radiology, Massachusetts General Hospital, Harvard Medical School

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers between 21 and 64 years of age with chronic pelvic pain for more than six months by self report. Six months of chronic pain is the criteria most often used in CPP research.
* CPP diagnoses will include endometriosis pain.
* Average pain intensity of ≥4 on a scale from 0 to 10, because <4 is considered a level with acceptable pain and function
* At least an 8th grade English-reading level; English can be a second language provided that the subjects feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Any interventional procedure for CPP two weeks prior to the study or during the two-week study period, such as lumbar epidural steroids, nerve root blocks, etc.
* Any etiology for CPP due to a known local somatic lesion for the pain (e.g. fibroids etc.) documented by the patient's gynecologist, surgery and/or imaging. We wish to focus on functional CPP, which may be more amenable to RAVANS due to the systemic nature of VNS.
* Opioid usage, either oral or intrathecal.
* Surgical therapy in the previous 12 weeks, the intent to undergo surgery during the study period, or any clinically unstable systemic illness that is judged to interfere with the trial.
* Non-ambulatory status
* History of cardiac or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome.
* An inability to complete questionnaires accurately.
* Cancer or other malignant disease, except carcinoma in situ of the skin
* Pregnancy

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Characterize analgesia following verum and sham RAVANS treatment in Endometriosis patients with and without psychiatric co-morbidity. | 2-3 weeks
  This will be done by comparing the quantitative sensory testing between the real and sham vagus nerve stimulation sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States